CLINICAL TRIAL: NCT00603070
Title: Electronic Prescribing and Electronic Transmission of Discharge Medication Lists to Improve Ambulatory Medication Safety
Brief Title: Electronic Prescribing and Electronic Transmission of Discharge Medication Lists
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); New York Presbyterian Hospital (Other); Columbia University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: R18HS017029-01 (AHRQ)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Medication Errors
Keywords: Medication Errors; Adverse Drug Events; Patient Safety; Electronic Prescribing Systems; Medication Reconciliation
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: All physicians and nurse practitioners at 1 ambulatory care clinics
  Interventions: Other: E-prescribing system
- 2: All physicians and nurse practitioners at 1 ambulatory care clinics
  Interventions: Other: Electronic transmission of medication discharge lists

INTERVENTIONS:
Other: E-prescribing system — Transition from home-grown to vendor-based ambulatory e-prescribing systems
  Other Names: WebCIS; CLIMACS; EpicCare; Eclypsis
  Groups: 1
Other: Electronic transmission of medication discharge lists — Patient discharge medication lists will be transmitted upon discharge from their inpatient medical record to their outpatient medical record and their outpatient provider will be notified of this transmission.
  Groups: 2

SUMMARY:
The purpose of this study is twofold:

1. to measure the effects of transitioning from one electronic prescribing system to another in the ambulatory setting on medication errors and human-computer interactions
2. to evaluate the impact of electronic transmission of discharge medication lists to the ambulatory setting on medication discrepancies and adverse drug events

ELIGIBILITY:
Inclusion Criteria:

* Physicians or nurse practitioners with at least 4 clinic sessions per week

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians and Nurse Practitioners from 2 office practices in the Ambulatory Care Network at NYPH, Associates in Internal Medicine (AIM) on the Columbia campus and Cornell Internal Medicine Associates (CIMA) on the Cornell campus.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Prescription medication errors | 2 weeks prior, 3 months, 1 year after intervention and 2 years after intervention
Medication discrepancies (as detected on a comparison between inpatient and outpatient medical records) | 30 days after patient is discharged from hospital
Patient adverse drug events (as determined by patient telephone interview and medical record review) | 30 days after patient hospital discharge

SECONDARY OUTCOMES:
Human-Computer interactions as measured by physician interview and direct observation of physician work | 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rainu Kaushal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Internal Medicine Associates, New York, New York, United States

REFERENCES:
- [Derived] Abramson EL, Malhotra S, Osorio SN, Edwards A, Cheriff A, Cole C, Kaushal R. A long-term follow-up evaluation of electronic health record prescribing safety. J Am Med Inform Assoc. 2013 Jun;20(e1):e52-8. doi: 10.1136/amiajnl-2012-001328. Epub 2013 Apr 11. PMID 23578816
- [Derived] Abramson EL, Patel V, Malhotra S, Pfoh ER, Nena Osorio S, Cheriff A, Cole CL, Bunce A, Ash J, Kaushal R. Physician experiences transitioning between an older versus newer electronic health record for electronic prescribing. Int J Med Inform. 2012 Aug;81(8):539-48. doi: 10.1016/j.ijmedinf.2012.02.010. Epub 2012 Mar 30. PMID 22465355
- [Derived] Abramson EL, Malhotra S, Fischer K, Edwards A, Pfoh ER, Osorio SN, Cheriff A, Kaushal R. Transitioning between electronic health records: effects on ambulatory prescribing safety. J Gen Intern Med. 2011 Aug;26(8):868-74. doi: 10.1007/s11606-011-1703-z. Epub 2011 Apr 16. PMID 21499828